CLINICAL TRIAL: NCT02472951
Title: Cut Down on Carbohydrate Usage in the Diet of Type 2 Diabetes - Mechanisms of Effective Therapy of Diabetes by Selective Choice of Macronutrients - The Phenotype Study
Acronym: CutDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Amirsalar Samkani, MD, PhD-stud, Bispebjerg Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 46559
Record Dates: First submitted 2015-06-12; First posted 2015-06-16 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Type 2 diabetic subjects (Active Comparator)
  Interventions: Other: Low carbohydrate meals; Other: Standard carbohydrate meals
- Prediabetic subjects (Active Comparator)
  Interventions: Other: Low carbohydrate meals; Other: Standard carbohydrate meals
- Healthy subjects (Active Comparator)
  Interventions: Other: Low carbohydrate meals; Other: Standard carbohydrate meals

INTERVENTIONS:
Other: Low carbohydrate meals — Meal macronutritional energy composition:
  Carbohydrate 30% Protein 30% Fat 40%
Other: Standard carbohydrate meals — Meal macronutritional energy composition:
  Carbohydrate 55% Protein 15% Fat 30%

SUMMARY:
Scientific evidence for the dietary treatment of type 2 diabetes is insufficient. The investigators hypothesize that a lower carbohydrate content in the diabetic diet than the recommended 55 E% will decrease the postprandial glucose excursion, decrease insulinotropic factors like incretin hormones and decrease their insulinotropic effects due to their glucose dependency. This will reduce postprandial insulin concentration, resulting in an improved insulin sensitivity and glucose metabolism. This clinical study will examine in diabetic, prediabetic and healthy subjects the acute effects of short term highly controlled dietary low carbohydrate intervention on metabolic pathways with respect to insulin action, pancreatic islet function, lipid metabolism, incretin hormones, low grade inflammation in plasma and novel measures of fatty acid metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Men age 18-70 years
* Postmenopausal women age 55-70 years
* Non-smoker (abstinent at least 6 months)
* HbA1c < 74 mmol/mol
* Fasting blood glucose < 11 mmol/L (mean of 3 measurements)
* Negative (<25 IU/L) plasma glutamate decarboxylase (GAD-65) antibodies (IgG)
* Hemoglobin > 7.5 mmol/L (men); > 6.8 mmol/L (women)
* Normal thrombocytes (140-400 x 109/L)
* eGFR > 45 ml/min per 1.73 m2
* Alkaline phosphatase < 140 IU/L
* Alanine aminotransferase < 70 IU/L
* Normal International Normalized Ratio (0.9-1.2)

Exclusion Criteria:

* Critical illness
* Anti-diabetic drugs other than metformin (maximum of 2000 mg / day)
* Steroid treatment e.g. prednisolone
* Reported or journalized severe food allergy or intolerance
* Reported or journalized gut disease e.g. Crohn's disease, Coeliac disease
* Reported or journalized alcohol dependence syndrome

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | Measured during meal tests (2 days with each intervention)
  Insulin sensitivity as measured by the oral minimal model applied to the meal test

CONTACTS AND LOCATIONS:
Overall Officials: Steen B Haugaard, MD, DMSc, associate prof., Study Director — Amager og Hvidovre Hospital; Thure Krarup, MD, DMSc, Study Director — Bispebjerg Hospital; Amirsalar Samkani, MD, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Endocrinological Dept. Bispebjerg University Hospital, Copenhagen, Region Sjælland, Denmark

REFERENCES:
- [Derived] Thomsen MN, Skytte MJ, Samkani A, Astrup A, Fenger M, Frystyk J, Hartmann B, Holst JJ, Larsen TM, Madsbad S, Magkos F, Rehfeld JF, Haugaard SB, Krarup T. Weight loss improves beta-cell function independently of dietary carbohydrate restriction in people with type 2 diabetes: A 6-week randomized controlled trial. Front Nutr. 2022 Aug 19;9:933118. doi: 10.3389/fnut.2022.933118. eCollection 2022. PMID 36061897
- [Derived] Thomsen MN, Skytte MJ, Astrup A, Deacon CF, Holst JJ, Madsbad S, Krarup T, Haugaard SB, Samkani A. The clinical effects of a carbohydrate-reduced high-protein diet on glycaemic variability in metformin-treated patients with type 2 diabetes mellitus: A randomised controlled study. Clin Nutr ESPEN. 2020 Oct;39:46-52. doi: 10.1016/j.clnesp.2020.07.002. Epub 2020 Aug 1. PMID 32859328
- [Derived] Samkani A, Skytte MJ, Anholm C, Astrup A, Deacon CF, Holst JJ, Madsbad S, Boston R, Krarup T, Haugaard SB. The acute effects of dietary carbohydrate reduction on postprandial responses of non-esterified fatty acids and triglycerides: a randomized trial. Lipids Health Dis. 2018 Dec 27;17(1):295. doi: 10.1186/s12944-018-0953-8. PMID 30591062
- [Derived] Samkani A, Skytte MJ, Kandel D, Kjaer S, Astrup A, Deacon CF, Holst JJ, Madsbad S, Rehfeld JF, Haugaard SB, Krarup T. A carbohydrate-reduced high-protein diet acutely decreases postprandial and diurnal glucose excursions in type 2 diabetes patients. Br J Nutr. 2018 Apr;119(8):910-917. doi: 10.1017/S0007114518000521. PMID 29644957